CLINICAL TRIAL: NCT06041776
Title: A Multicenter, Randomized, Controlled, Double Blind, Double Simulated, Phase III Clinical Study of Befotertinib vs Icotinib for Postoperative Adjuvant Treatment of IB-IIIB (T3N2M0) Stage Non Small Cell Lung Cancer With Positive EGFR Sensitive Mutations
Brief Title: Adjuvant Befotertinib in Stage IB-IIIB Non-small Cell Lung Cancer With Positive EGFR Sensitive Mutations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BD-BF-III01
Record Dates: First submitted 2023-09-12; First posted 2023-09-18 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Non-Small Cell Lung Cancer; EGFR Sensitive Mutation; Adjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Befotertinib + Icotinib placebo (Experimental): Befotertinib (75 mg or 100 mg orally, once daily) and Icotinib placebo(125 mg orally, three times daily)，in accordance with the randomization schedule
  Interventions: Drug: Befotertinib + Icotinib placebo
- Icotinib + Befotertinib placebo (Active Comparator): Icotinib (125 mg orally, three times daily) and Befotertinib placebo (75 mg or 100 mg orally, once daily)，in accordance with the randomization schedule
  Interventions: Drug: Icotinib + Befotertinib placebo

INTERVENTIONS:
Drug: Befotertinib + Icotinib placebo — The initial dose of Befotertinib is 75 mg orally once daily (QD) for 21 days, and then increased to 100 mg orally QD in the absence of serious side effects , CTCAE grade ≥ 2 headache or thrombocytopenia during the 21 days.
  Befotertinib can be taken on an empty stomach or after meals, and the medication is used until the disease relapses or intolerable toxicity occurs, or the treatment lasts for 3 years (disease recurrence includes local recurrence and/or distant metastasis)
  Icotinib placebo 125 mg three times daily, on an empty stomach or in combination with food, use medication until the disease relapses or intolerable toxicity occurs or treatment lasts for 2 years (disease recurrence includes local recurrence and/or distant metastasis).
  Arms: Befotertinib + Icotinib placebo
Drug: Icotinib + Befotertinib placebo — Icotinib 125 mg three times daily, on an empty stomach or in combination with food, use medication until the disease relapses or intolerable toxicity occurs or treatment lasts for 2 years (disease recurrence includes local recurrence and/or distant metastasis).
  The initial dose of Befotertinib placebo is 75 mg orally once daily (QD) for 21 days, and then increased to 100 mg orally QD in the absence of serious side effects , CTCAE grade ≥ 2 headache or thrombocytopenia during the 21 days.
  Befotertinib placebo can be taken on an empty stomach or after meals, and the medication is used until the disease relapses or intolerable toxicity occurs, or the treatment lasts for 3 years (disease recurrence includes local recurrence and/or distant metastasis.
  Arms: Icotinib + Befotertinib placebo

SUMMARY:
This multicenter, randomized, controlled, double-blind, double-simulated, Phase III study is designed to evaluate the efficacy and safety of Befotertinib compared with Icotinib as adjuvant treatment in EGFR-sensitive mutation-positive stage IB-IIIB (T3N2M0) non-small cell lung cancer after surgical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to sign informed consent prior to any study specific procedures, and ability to with scheduled visits, treatment plans, laboratory tests, and other study procedures.
2. Male or female, aged at least 18 years.
3. Histologically confirmed primary NSCLC, and mainly non-squamous cell carcinoma (including mixed type carcinoma mainly composed of adenocarcinoma components).
4. Absence of brain metastasis.
5. Complete resection of histologically confirmed Stage IB, II, IIIA or IIIB(T3N2M0) according to the TNM staging system for lung cancer (AJCC/UICC 8th edition), with negative margins.
6. Confirmation by the central laboratory that the tumor harbors one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R).
7. Patients who fully recover from surgery during randomization (any surgery must achieve complete postoperative wound healing) and should receive adjuvant treatment within 4-10 weeks after surgery.
8. ECOG-PS score of 0 or 1 and did not deteriorate 2 weeks before the first administration of the investigational drug, with a minimum expected survival greater than 12 weeks.
9. Female subjects with fertility need to have a negative serum pregnancy test during screening.
10. Female subjects who have possibility of becoming pregnant, as well as male subjects whose partners are women of childbearing age, must use a highly effective contraceptive method (such as oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicides) throughout the study and continue to use contraception for 3 months after the end of treatment.

Exclusion Criteria:

1. There are unresectable or metastatic diseases, pathological reports showing positive surgical margins under the microscope or extranodal invasion, or lesions left after surgery, or suspicious lesions determined by imaging after surgery. Subjects receiving only wedge resection.
2. Upper lung groove cancer.
3. Patient with complete resection of the right lung with NSCLC.
4. Malignancies other than NSCLC within 5 years prior to first dosage, except for malignant tumors that can be cured after treatment (including but not limited to fully treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or breast ductal carcinoma in situ treated with radical surgery).
5. Received systematic anti-tumor therapy, including chemotherapy, radiotherapy or targeted therapy (including but not limited to monoclonal antibodies, small molecule tyrosine kinase inhibitors), immunotherapy, investigational therapy, etc., before being enrolled in this study.
6. Within 3 weeks prior to the first administration of the investigational drug, the patient underwent major surgery (including primary tumor surgery, craniotomy, thoracotomy, or laparotomy, excluding vascular pathway establishment procedures).
7. Within 14 days prior to first dose of the investigational drug, Traditional Chinese medicine with anti-tumor indications have been received.
8. After the start of the study, any form of systemic or local anti-tumor treatment (including maintenance therapy with another drug, radiotherapy, and/or surgical resection) is still required.
9. Clinically significant cardiovascular diseases, including:

   1. QTcF interval >450 ms (men) or >470 ms (women), symptomatic bradycardia (<45 beats /min), or other significant ECG abnormalities as determined by the investigator (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec).
   2. Echocardiography showed LVEF <50%.
   3. Hypertension was clinically uncontrollable (e.g., blood pressure >160/100 mmHg; Except that isolated elevated readings that were determined by the investigators to be clinically insignificant or controllable hypertension.)

   Within 6 months before the first medication, there were the following situations:
   1. Congestive heart failure (New York Heart Association rating III or IV).
   2. Arrhythmias or conduction abnormalities that require medication treatment. Note: Patients with drug-controlled atrial fibrillation/flutter, as well as those with pacemaker- controlled arrhythmia, can be selected.
   3. Severe/unstable angina, coronary artery/peripheral bypass grafting, or myocardial infarction (Note: Severe angina is classified as Grade III or IV by the Canadian Society of Cardiology).
   4. Cerebrovascular accidents or transient ischemic attacks, transient myocardial ischemia.
10. Previous history of concomitant interstitial lung disease (ILD), drug-induced ILD, radiation pneumonia requiring hormone therapy, or clinical evidence of concomitant active interstitial lung disease.
11. Patients who have a history of thrombosis or are currently present with thrombosis or have a potential risk of thrombosis assessed by the investigator.
12. Any clinical evidence of a serious active infection, or any serious concomitant disease that may affect the subject's acceptance of investigational drugs, such as active bleeding predisposition, active hepatitis B, hepatitis C, or tuberculosis, syphilis, or HIV antibody positive.
13. There are serious gastrointestinal functional abnormalities in clinical practice that may affect drug intake, transportation, or absorption, such as inability to take medication orally, uncontrollable nausea or vomiting, history of extensive gastrointestinal resection, untreated recurrent diarrhea, atrophic gastritis, untreated stomach diseases requiring long-term use of proton pump inhibitors, gastrointestinal obstruction, active diverticulitis, Crohn's disease, ulcerative colitis, etc.
14. Abnormal laboratory parameters.
15. Known hypersensitivity to the befotertinib, icotinib or their inactive excipients.
16. Within one week before the first administration of the investigational drug, it is currently in use or needs to be combined with CYP3A strong inhibitors or inducers during the study period.
17. Patients who are still using warfarin within 7 days prior to initial dosing (low molecular weight heparin sodium is allowed).
18. Participating in clinical research and receiving treatment with the study drug or research device, or participating in clinical research and receiving treatment with the study drug or research device within 4 weeks before the first administration, or planning to participate in any other clinical trial during this study period.
19. Inoculate with a live vaccine within 180 days before the first medication.
20. Researchers believe that it may affect protocol compliance or affect the signing of informed consent forms by participants (such as a history of mental illness or drug abuse, alcoholism or other addiction), or any other clinically significant disease or condition that is not suitable for participation in this clinical trial (such as laboratory abnormal results, clinically active diverticulitis, abdominal abscess).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) evaluated by investigator in patients with stage II-IIIB (T3N2M0) | up to 5 years

SECONDARY OUTCOMES:
DFS evaluated by investigator in patients with stage IB-IIIB (T3N2M0) | up to 5 years

OTHER OUTCOMES:
DFS rate at 2 years | Assessed at 2 years
DFS rate at 3 years | Assessed at 3 years
DFS rate at 5 years | Assessed at 5 years
Overall survival (OS) | Assessed at 5 years
OS rate at 5 years | up to 5 years
Treatment-Emergent Adverse Event (TEAE) | Until 28 days after the last dosing

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, M.D., Study Chair — Shanghai Chest Hospital
Locations (3):
- China (3):
  - Peking University International Hospital, Beijing
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai chest hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No